CLINICAL TRIAL: NCT00471770
Title: Epidemiological Study of Hospitalized Pediatric Pneumonia in China
Brief Title: Pneumoniae Epidemiology Study in China
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0887X-101894
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — deep respiratory aspirate,pleural fluid,cerebrospinal fluid,serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: 1.Core group: enrolled subjects who have isolated pneumococcal
- 2: 2.SPN group:enrolled subjects who have no isolated pneumococcal
- 3: 3.DCF group: Subjects screened but not enrolled

SUMMARY:
To determine the proportion of hospitalized pneumonia cases in children aged 60 months or less associated with vaccine-preventable Streptococcus pneumoniae serotypes (4, 6B, 9V, 14, 18C, 19F, 23F).

DETAILED DESCRIPTION:
Subjects meeting the eligibility criteria, including parental informed consent to collect clinical-epidemiological information, will have a deep respiratory aspirate specimen to determine the etiology of the lower respiratory tract infection. Clinicians may obtain other diagnostic specimens, such as pleural fluid, lung tap, cerebrospinal fluid, nasopharyngeal culture, or serum for serological assays, as indicated clinically. The chest radiograph will be taken and read locally according to predetermined criteria and by staff radiologists trained in radiographic criteria for pneumonia. Bacterial isolates other than Streptococcus pneumoniae will be identified according to standardized procedures. S. pneumoniae isolates will be transported to central laboratories for confirmation of identity, serotyping and antibiotic resistance testing, using standard techniques. Serotype will be determined using type-specific sera (Quellung reaction). Antibiotic susceptibility to penicillin, cefuroxime, ceftriaxone, erythromycin, Amoxycillin, Ofloxacin, Vancomycin, and imipenem be conducted using E-test according to standardized procedures at the central facilities.

ELIGIBILITY:
Inclusion Criteria:

* Age, 60 months or less
* Meets study criteria for clinical pneumonia
* All the examination are/can be done within (before or after) 72 hours to enrollment time
* Informed consent obtained from parent or guardian

Exclusion Criteria:

* Received any pneumococcal vaccine in the past
* Current or underlying conditions that would pose a hazard in obtaining the deep respiratory aspirate (e.g., bleeding diathesis, severe respiratory compromise and others as determined by clinician) Aspirates may be obtained from patients who are intubated
* Any other medical condition that in the opinion of the clinician/investigator would pose a hazard to the child by participating in the study
* Children with recurrent pneumonia will enter into the study on only one occasion

Max Age: 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalized children with pneumoniae less than 5 years,located in Tianjin Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The proportion of hospitalized pneumonia cases associated with vaccine-preventable S. Pneumoniae serotypes (4, 6B, 9V, 14, 18C, 19F, 23F). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tianjin, China